CLINICAL TRIAL: NCT01743157
Title: A Phase I-II Study of Treatment of Metastatic Melanoma Using Induction Therapy With Biochemotherapy and Bevacizumab Followed by Consolidation Therapy With Ipilimumab (BBI)
Brief Title: Biochemotherapy and Bevacizumab Followed by Consolidation Therapy With Ipilimumab for Metastatic Melanoma
Acronym: BBI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: Principal Investigator, David Minor, MD, Medical Doctor, California Pacific Medical Center Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBI Total Therapy
Expanded Access: NCT00495066 (No longer available)
Record Dates: First submitted 2011-04-04; First posted 2012-12-06 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab; Temozolomide; Cisplatin; Vinblastine; Interleukin-2; Introns; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biochemo + Bevacizumab then Ipilimumab (Experimental): Single arm: Biochemotherapy with 4 cycles at 3 week intervals of Temozolamide 150mg/m2 x4, cisplatin 20mg/m2 x 4, vinblastine 1.2mg/m2 x 4, bevacizumab 7.5-15 mg/kg x 1, interferon 5mg/m2 x5 and aldesleukin 36,18,9, % 9 miu/day over 4 days each cycle; then ipilimumab 3mg/kg q 21 days x 4, then q 3 months x 8 for total 3 years.
  Interventions: Drug: Biochemo + bevacizumab then ipilimumab

INTERVENTIONS:
Drug: Biochemo + bevacizumab then ipilimumab — Bevacizumab 7.5mg/kg week 1,repeat weeks 4,7,10 (cycles 2, 3, & 4)
  Other Names: Avastin,; Temodar,; Platinol,; Velban,; interleukin-2,; Intron-A,; Yervoy

SUMMARY:
A phase I-II study of treatment of metastatic melanoma using induction therapy with Biochemotherapy plus Bevacizumab followed by consolidation therapy with Ipilimumab (BBI).

DETAILED DESCRIPTION:
A phase I-II study of treatment of metastatic melanoma using induction therapy with Biochemotherapy (Temodar,Cisplatin, Velban,IL2 and IFN)plus Bevacizumab followed by consolidation therapy with Ipilimumab (BBI)

ELIGIBILITY:
Inclusion Criteria:

1. Stage 4 or unresectable stage 3 metastatic melanoma with or without measurable disease
2. Age 18-70 years old
3. Adequate pulmonary and cardiac function for high-dose IL-2
4. PS 0-2
5. Previous ipilimumab therapy will not exclude patients, but patients with previous ipilimumab will have separate efficacy analysis

Exclusion Criteria:

1. Brain metastases
2. Creatinine > 2x ULN; bilirubin > 3, WBC < 3500, Platelets < 100,000, Hgb < 9
3. Another active malignancy
4. Gastrointestinal tract metastases except rectal metastases or primary are allowable
5. Previous therapy for metastatic disease with chemotherapy of duration over 3 months or with high-dose interleukin-2
6. History of colitis or autoimmune disease such as lupus or rheumatoid arthritis
7. Bevacizumab-related contraindications: Hemoptysis or history of severe bleeding, uncontrolled hypertension, proteinuria with protein/creatinine ratio > 1, acute myocardial infarction within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
A phase I-II study of treatment of metastatic melanoma using induction therapy with Biochemotherapy and Bevacizumab followed by consolidation therapy with Ipilimumab (BBI) | Primary Objective
  Determine the incidence of grade 4 bevacizumab-related toxicities and grade 3 proteinuria when bevacizumab is given with biochemotherapy to patients with metastatic melanoma for up to 3 years.

SECONDARY OUTCOMES:
A phase I-II study of treatment of metastatic melanoma using induction therapy with Biochemotherapy and Bevacizumab followed by consolidation therapy with Ipilimumab (BBI) | Secondary Objective
  Compare median and overall progression-free survival to previously published historical control group of 135 patients receiving biochemotherapy followed by pulse IL-2, and also patients in the study of Weber et al (Reference 9) of ipilimumab in previously untreated patients for up to 4 years.

CONTACTS AND LOCATIONS:
Overall Officials: David R Minor, MD, Principal Investigator — California Pacific Medical Center
Locations (1):
- San Francisco Oncology Associates, San Francisco, California, United States

REFERENCES:
- [Result] 3. Minor DR, Wang W, Kashani-Sabet: Concurrent bevacizumab (BEV) with biochemotherapy (BIO) followed by ipilimumab for advanced melanoma: a phase I-II trial. J Clin Onc 2013 (suppl; abstr e200001)